CLINICAL TRIAL: NCT04084977
Title: Sydenham's Chorea: Is There a Link Between Neuropsychiatric Symptoms and Anti-dopamine Receptor Autoantibodies?
Brief Title: Dopaminergic Receptors in Sydenham's Chorea
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 139/14
Record Dates: First submitted 2019-01-02; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Sydenham Chorea; Strep Throat
MeSH Terms: conditions — Chorea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Sera
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sydenam Chorea (SC): individuals with SC
  Interventions: Diagnostic Test: Antibody detection
- tonsilitis: children with tonsilitis in the past 3 months
  Interventions: Diagnostic Test: Antibody detection
- control: children wit no tonsilitis
  Interventions: Diagnostic Test: Antibody detection

INTERVENTIONS:
Diagnostic Test: Antibody detection — detecting anti bodies against D1, D2 receptor, tubolin Lysoganglioside

SUMMARY:
Sydenham's chorea (SC) is a post-streptococcal, neuropsychiatric disorder associated with anti-neuronal antibodies. The investigators demonstrated elevated anti-D1-receptor (D1R) and anti-D2-receptor (D2R) antibodies titers compared to controls using ELISA. Similarly, the investigators found antibodies to surface D2R in neuropsychiatric, autoimmune disorders, including SC using cell-based assays. The investigators hypothesize that these autoantibodies cause neuropsychiatric symptoms by inducing intracellular signaling changes resulting in altered dopaminergic neurotransmission. To check this, the investigators will test whether sera from patients with SC alter dopaminergic signaling pathways. The investigators will examine sera from 30 SC patients with active symptoms and 30 age-matched healthy controls. Patients with SC will be assessed for severity of neuropsychiatric symptoms using UFMG Sydenham's Chorea Rating Scale. Controls with evidence of streptococcal infections or autoimmune disorders will be excluded. Sera will be examined for anti-D1R and anti-D2R antibodies. Signaling studies will assess sera impact on 1) calcium/calmodulin-dependent protein kinase II activity in human neuronal cells. 2) dopamine D1/D2 receptors signaling using cAMP assays in transfected cell lines. The investigators will examine the correlation between modified signaling and clinical symptoms.

DETAILED DESCRIPTION:
Participants:

The investigators will enroll participants with acute Sydenham's chorea (aSC) and age-matched controls with streptococcal tonsillitis (ST) within the past 4 months and healthy children (HC) with no a history of a strep infection in the past 6 months and negative throat culture. Informed consent will be obtained from participants and/ or parents. Children with SC will be evaluated for SC severity using the USCRS. The investigators will record clinical data regarding gender, age, duration symptoms, and medical treatments. Controls will be examined by referring physician to rule out chorea. Sera samples from all participants will be stored at -70°C and shipped to the microbiology and immunology lab, University of Oklahoma Health Sciences Center (OHSC) on dry ice.

Laboratory testing:

Immunophenotyping for anti-D1R, anti-D2R, anti- LG and anti-tubulin titers and signaling studies will be performed at the OUHSC microbiology and immunology laboratory.

Autoantibody titers. Sera will be assayed for reactivity with the dopamine D1 and D2 receptors (Human dopamine D1 and D2 receptor membrane antigens, Perkin Elmer-Membrane Target Systems) in the direct ELISA and assays which include the ELISA competitive inhibition. Anti- LG and anti-tubulin titers will be tested as well.

Statistical Analysis:

Time will be categorized in order to model non-linear associations among the groups. Means will be compared among groups using an ANOVA model that included main effects for the time, participant diagnosis and the interaction between participant diagnosis and time. Modeling assumptions will be evaluated using residual plots. A natural log transformation of the antibody measure will be used when there was evidence of non-constant variance across the groups. If a significant interaction between time and participant group will be found, time trends will be summarized separately within each participant group. Post-hoc pair-wise comparisons will be made using Tukey's method to control the type I error rate. A two-sided 0.05 alpha level will be used to define statistical significance. Analyses will be performed using SAS (SAS Institute Inc., SAS v9.4, Cary, NC: SAS Institute Inc.).

ELIGIBILITY:
Inclusion Criteria:

* sydenham chora OR strep tonsilitiscontrol without strep tonsilitis OR

Exclusion Criteria:

* neurological disrder autoimmune disorder

Ages: 2 Years to 40 Years | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: sydenhams chorea according to clinical parameters
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Antibody titers | Once at time of initial visit within the first 4 months from onset
  titer levels of anti dopamine receptors (anti-D1 and anti-D2) using ELISA (titer levels are expresed as dilutions i.e. 1:400)
UFMG Sydenham's Chorea Rating Scale | Upon presentation when symptomatic, usually within 4 months of onset
  the mean value of the 21 item of clinical chorea rating. Ranging from 0 (=none) to 4 (=severe) for each item

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical center, Jerusalem, Israel